CLINICAL TRIAL: NCT01907152
Title: Increase Protein Intake in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Fonterra (Europe) Cooperatie U.A. (Unknown); Carezzo B.V. (Other); Amsterdam UMC, location VUmc (Other); Hogeschool van Arnhem en Nijmegen (HAN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL43997.081.13; TKI-AF 12065 (Other Grant/Funding Number: Stichting Topconsortium voor Kennis en Innovatie Agri & Food)
Record Dates: First submitted 2013-07-22; First posted 2013-07-24 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Markedly Reduced Food Intake
Keywords: malnutrition; undernourishment; loss of muscle mass
MeSH Terms: conditions — Malnutrition | interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein enriched yoghurt drink and bread (Experimental): Yoghurt drink enriched with Whey Protein Concentrate Whole wheat bread enriched with cereal protein and soy
  Interventions: Other: Protein enriched yoghurt drink and bread
- Regular yoghurt drink and bread (No Intervention): Commercially available yoghurt drink and whole wheat bread

INTERVENTIONS:
Other: Protein enriched yoghurt drink and bread
  Arms: Protein enriched yoghurt drink and bread

SUMMARY:
The objective of this study is to investigate the acceptance, intake, and compliance of protein enriched bread and protein enriched yoghurt drinks in elderly patients in two real life settings (short term; hospital, and longer term; rehabilitation home).

DETAILED DESCRIPTION:
Prevalence rates of protein-energy malnutrition in elderly are high. In order to prevent loss of muscle mass and remain physically independent, it is utmost important for elderly to maintain their body protein mass. A sufficient protein supply according to their needs is therefore highly important. Especially for frail elderly, it is not easy to realize an increased protein intake by simply eating more. It is hypothesized that protein enriched food products that fit in a habitual diet (dairy and bread), result in a higher protein intake compared to regular products.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the department of internal medicine of VU university medical center or to the rehabilitation department of "Herstelhotel Dekkerswald"
* signed informed consent
* age of 55 or more
* rehabilitating from a hospital stay with the aim to return back home (rehabilitation home only)
* likely to remain admitted at least 3 weeks (rehabilitation home only).

Exclusion Criteria:

* not speaking Dutch language
* allergy for milk, soy or gluten
* a medical condition that is considered by the treating physician as a contra indication for receiving protein enriched food products
* a diet that does not allow the use of normal bread or dairy products (e.g. fluid diet, strong sodium restricted diet)
* not able to eat or feed themselves
* receiving tube feeding or parenteral nutrition
* suffering from a terminal illness

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Protein intake measured on an individual level over 24h | 3 days (hospital), 3 weeks (rehabilitation home)

SECONDARY OUTCOMES:
Intake of macronutrients (besides protein), total energy, calcium and fibre measured on an individual level over 24h. | 3 days (hospital), 3 weeks (rehabilitation home)

OTHER OUTCOMES:
Product evaluation | 3 days (hospital), 3 weeks (rehabilitation home)
  Questionnaire on appreciation and acceptance of protein enriched food products

CONTACTS AND LOCATIONS:
Overall Officials: Esther Boelsma, PhD, Principal Investigator — Wageningen UR Food and Biobased Research
Locations (2):
- Netherlands (2):
  - VU university medical center, Amsterdam
  - Rehabilitation home "Herstelhotel Dekkerswald", Groesbeek

REFERENCES:
- [Derived] Stelten S, Dekker IM, Ronday EM, Thijs A, Boelsma E, Peppelenbos HW, de van der Schueren MA. Protein-enriched 'regular products' and their effect on protein intake in acute hospitalized older adults; a randomized controlled trial. Clin Nutr. 2015 Jun;34(3):409-14. doi: 10.1016/j.clnu.2014.08.007. Epub 2014 Aug 15. PMID 25179468